CLINICAL TRIAL: NCT05470673
Title: The Effect of Autogenous Demineralized Dentin Graft Combined With Injectable PRF Loaded With Metronidazole Versus Autogenous Demineralized Dentin Graft Alone on Alveolar Ridge Preservation of Infected Sockets: A Randomized Controlled Clinical Trial
Brief Title: Autogenous Demineralized Dentin Graft Combined With Injectable PRF + Metronidazole Versus Autogenous Demineralized Dentin Graft Alone for Alveolar Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Talaat Mohamed Mahmoud El Behwashy, Principal Investigator. Mohamed Elbehwashy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: perio2022ARP
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar ridge preservation using demineralized dentin combined with I-PRF + metronidazole (Experimental): Atraumatic extraction of non-restorable teeth, then the extracted tooth will be prepared and demineralized using hydrochloric acid (HCL) acid as particulate demineralized dentin graft and processed with injectable platelet rich fibrin. The injectable PRF will be mixed with 5mg/ml metronidazole first then added to the particulate demineralized dentin graft then inserted in the extraction socket and covered then suturing
  Interventions: Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft combined with injectable PRF loaded with metronidazole
- Alveolar ridge preservation using autogenous demineralized dentin graft alone (Active Comparator): Atraumatic extraction of non-restorable teeth, then the extracted tooth will be prepared and demineralized using hydrochloric acid (HCL) acid as particulate demineralized dentin graft and inserted in the extraction socket and covered then suturing
  Interventions: Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft alone

INTERVENTIONS:
Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft combined with injectable PRF loaded with metronidazole — Atraumatic extraction of non-restorable teeth, then the extracted tooth will be prepared and demineralized using hydrochloric acid (HCL) acid as particulate demineralized dentin graft and processed with injectable platelet rich fibrin. The injectable PRF will be mixed with 5mg/ml metronidazole first then added to the particulate demineralized dentin graft forming sticky demineralized tooth graft with slowly released metronidazole then inserted in the extraction socket and covered then suturing
  Arms: Alveolar ridge preservation using demineralized dentin combined with I-PRF + metronidazole
Procedure: Alveolar ridge preservation using autogenous demineralized dentin graft alone — Atraumatic extraction of non-restorable teeth, then the extracted tooth will be prepared and demineralized using hydrochloric acid (HCL) acid inserted in the extraction socket as particulate demineralized dentin graft
  Arms: Alveolar ridge preservation using autogenous demineralized dentin graft alone

SUMMARY:
The aim of this trial is to compare the effect of autogenous demineralized dentin graft combined with injectable PRF loaded with metronidazole (sticky demineralized tooth releasing metronidazole) versus autogenous demineralized dentin graft (ADDG) alone on alveolar ridge preservation after extraction of non restorable, infected single-rooted teeth

DETAILED DESCRIPTION:
Many studies have reported an approximately 50% reduction in alveolar bone both the horizontal and vertical directions over 12 months with more than two-thirds of the reduction occurring in the first three months after extraction. Alveolar ridge preservation is a procedure that attempts to reduce bone dimensional changes that naturally take place following tooth extraction. During the last decade, efforts have been made to confirm procedures that can prevent bone resorption after extraction. The use of bone grafts aim to promote bone healing and assist bone regeneration. Various types of materials are used for socket preservation, such as autogenous bone, allograft bone, xenograft materials, and alloplast materials.

Dentin contains several growth factors, including transforming growth factor beta (TGF-β), insulin-like growth factor-II (IGF-II) and bone morphogenetic protein-2 (BMP-2), which could be of pivotal importance during any healing event. Demineralization of dentin has been further proposed to expose its collagen matrix, liberate 'fossilized' growth factors and thereby enhance its regenerative capacity.

It has been proven that autogenous demineralized dentin graft is effective at reducing dimensional losses of alveolar sockets after 6 months, with no adverse effects.

The efficacy of platelet rich fibrin (PRF) in promoting wound healing and tissue regeneration is at the center of a recent academic debate. The liquid fibrinogen has been shown to bind particulate bone grafts, which are then called "sticky bone". This binding improves the stabilization of the particles in the defect. It adds a potential biological effect, which could accelerate the soft tissue healing process and optimize the handling properties of the granules.

The purpose of this clinical trial is to assess the capacity and the clinical feasibility of the dentin graft processed with injectable platelet rich fibrin (I-PRF) to an adherent, tooth-derived conglomerate for socket preservation. Moreover, Platelet-rich fibrin incorporated with antibiotics showed long-term anti-bacterial effect against F. nucleatum and S. aureus.

Both autogenous demineralized dentin graft combined with injectable PRF (sticky demineralized tooth) and autogenous demineralized dentin graft (ADDG) alone, with or without collagen membrane, have been utilized for alveolar ridge preservation or augmentation but the superiority of one form over the other is not yet clear.

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable tooth indicated for extraction
* Single-rooted teeth
* Inactive infection related to the tooth
* Motivated patients, agree to sign informed consent and complete the follow-up period

Exclusion Criteria:

* Pregnant females
* Active infection at extraction site
* Smokers
* Systemic conditions affecting healing (e.g. diabetes, medications as bisphosphonates...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge apico-coronal height change in mm | 6 months
  Difference in height linear measurements between baseline and final CBCT scans

SECONDARY OUTCOMES:
Alveolar ridge bucco-lingual width change in mm | 6 months
  Alveolar bone linear width will be measured at baseline and after 6 months using cone beam computed tomography (CBCT) scans. The change in bone width will be calculated as the subtraction of final width from baseline width and will be measured in millimetres
Histological assessment | 6 months
  Bone samples from control and experimental sites will be taken during implant placement using a trephine bur of a size smaller than the implant. Samples will be examined for new bone formation (Yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Elfana A, El-Kholy S, Saleh HA, Fawzy El-Sayed K. Alveolar ridge preservation using autogenous whole-tooth versus demineralized dentin grafts: A randomized controlled clinical trial. Clin Oral Implants Res. 2021 May;32(5):539-548. doi: 10.1111/clr.13722. Epub 2021 Mar 1. PMID 33565656
- [Background] van Orten A, Goetz W, Bilhan H. Tooth-Derived Granules in Combination with Platelet-Rich Fibrin ("Sticky Tooth") in Socket Preservation: A Histological Evaluation. Dent J (Basel). 2022 Feb 16;10(2):29. doi: 10.3390/dj10020029. PMID 35200254